CLINICAL TRIAL: NCT06200103
Title: Minority-Inclusive Imaging Biomarker-Based End of Therapy Trial for 177Lu-PSMA-617, a Randomized De-Escalation Theranostic Trial for Metastatic Castrate Resistant Prostate Cancer
Brief Title: Schedule De-Escalation of 177Lu-PSMA-617 for the Treatment of Metastatic Castrate Resistant Prostate Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MC231005; NCI-2023-10664 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC231005 (Other: Mayo Clinic); MI-BET (Other: Mayo Clinic); 23-006547 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2023-12-28; First posted 2024-01-10 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Castration-Resistant Prostate Carcinoma; Stage IVB Prostate Cancer AJCC v8
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Specimen Handling; Watchful Waiting; Observation; gallium 68 PSMA-11; 68Ga-DKFZ-PSMA-11; Pluvicto; Magnetic Resonance Spectroscopy; X-Rays; Photons

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm I (177Lu-PSMA-617 standard) (Active Comparator): Patients receive 177Lu-PSMA-617 IV over 10-15 minutes on day 1 of each cycle. Cycles repeat every 42 days for 5 cycles in the absence of disease progression or unacceptable toxicity. Patients with a near complete response may receive 1 additional cycle. Patients receive gallium Ga 68-labeled PSMA-11 IV and undergo PET/CT and a bone scan during screening and on the trial. Patients also undergo SPECT/CT and blood sample collection on the trial.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Scan; Procedure: Computed Tomography; Other: Gallium Ga 68 Gozetotide; Drug: Lutetium Lu 177 Vipivotide Tetraxetan; Procedure: Positron Emission Tomography; Other: Questionnaire Administration; Procedure: Single Photon Emission Computed Tomography
- Arm II (177Lu-PSMA-617 treatment pause) (Experimental): Patients receive 177Lu-PSMA-617 IV over 10-15 minutes on day 1 of each cycle. Cycles repeat every 42 days for 5 cycles in the absence of disease progression or unacceptable toxicity. Patients then undergo clinical observation until documented first progression. After progression, patients resume treatment with 77Lu-PSMA-617 for another cycle. Patients receive gallium Ga 68-labeled PSMA-11 IV and undergo PET/CT and a bone scan during screening and on the trial. Patients also undergo SPECT/CT and blood sample collection on the trial.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Scan; Other: Clinical Observation; Procedure: Computed Tomography; Other: Gallium Ga 68 Gozetotide; Drug: Lutetium Lu 177 Vipivotide Tetraxetan; Procedure: Positron Emission Tomography; Other: Questionnaire Administration; Procedure: Single Photon Emission Computed Tomography
- Arm III (Treatment pause 177Lu-PSMA-617) (Experimental): Patients undergo clinical observation until documented first progression. After progression, patients receive 177Lu-PSMA-617 IV over 10-15 minutes on day 1 of each cycle. Cycles repeat every 42 days for 6 cycles in the absence of disease progression or unacceptable toxicity. Patients receive gallium Ga 68-labeled PSMA-11 IV and undergo PET/CT and a bone scan during screening and on the trial. Patients also undergo SPECT/CT and blood sample collection on the trial.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Scan; Other: Clinical Observation; Procedure: Computed Tomography; Other: Gallium Ga 68 Gozetotide; Drug: Lutetium Lu 177 Vipivotide Tetraxetan; Procedure: Positron Emission Tomography; Other: Questionnaire Administration; Procedure: Single Photon Emission Computed Tomography

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Scan — Undergo bone scan
  Other Names: Bone Scintigraphy
Other: Clinical Observation — Undergo active monitoring
  Other Names: observation
  Arms: Arm II (177Lu-PSMA-617 treatment pause); Arm III (Treatment pause 177Lu-PSMA-617)
Procedure: Computed Tomography — Undergo SPECT/CT or PET/CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; CT; CT Scan; tomography; Computerized Tomography (CT) scan
Other: Gallium Ga 68 Gozetotide — Given IV
  Other Names: (68)Ga labeled Glu-NH-CO-NH-Lys(Ahx)-HBED-CC; (68)Ga-labeled Glu-urea-Lys(Ahx)-HBED-CC; (68)Ga-PSMA Ligand Glu-urea-Lys(Ahx)-HBED-CC; (68)Gallium-PSMA Ligand Glu-urea-Lys(Ahx)-HBED-CC; (68Ga)Glu-urea-Lys(Ahx)-HBED-CC; 68Ga-DKFZ-PSMA-11; 68Ga-HBED-CC-PSMA; 68Ga-labeled Glu-NH-CO-NH-Lys(Ahx)-HBED-CC; 68Ga-PSMA; 68Ga-PSMA-11; 68Ga-PSMA-HBED-CC; [68Ga] Prostate-specific Membrane Antigen 11; [68Ga]GaPSMA-11; AAA 517; AAA-517; AAA517; Ga PSMA; Ga-68 labeled DKFZ-PSMA-11; Ga-68 labeled PSMA-11; GA-68 PSMA-11; Gallium Ga 68 PSMA-11; Gallium Ga 68-labeled PSMA-11; GALLIUM GA-68 GOZETOTIDE; Gallium-68 PSMA; Gallium-68 PSMA Ligand Glu-urea-Lys(Ahx)-HBED-CC; GaPSMA; PSMA-HBED-CC GA-68
Drug: Lutetium Lu 177 Vipivotide Tetraxetan — Given IV
  Other Names: 177Lu-labeled PSMA-617; 177Lu-PSMA-617; AAA 617; AAA-617; AAA617; Lu177-PSMA-617; Lutetium Lu 177-PSMA-617; LUTETIUM LU-177 VIPIVOTIDE TETRAXETAN; Lutetium-177-PSMA-617; Pluvicto
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging; PT
Other: Questionnaire Administration — Ancillary studies
Procedure: Single Photon Emission Computed Tomography — Undergo SPECT/CT
  Other Names: Medical Imaging, Single Photon Emission Computed Tomography; Single Photon Emission Tomography; Single-Photon Emission Computed; single-photon emission computed tomography; SPECT; SPECT imaging; SPECT SCAN; SPET; ST; tomography, emission computed, single photon; Tomography, Emission-Computed, Single-Photon

SUMMARY:
This phase II trial studies how to improve the usage of Lu 177 vipivotide tetraxetan (177Lu-prostate-specific membrane antigen [PSMA]-617) for treating patients with castration-resistant prostate cancer that has spread from where it first started (primary site), to other places in the body (metastatic) utilizing a treatment pause after 5 cycles of therapy versus standard continuous treatment for 6 cycles. Lutetium is a radioligand therapy (RLT). RLT uses a small molecule (in this case 177Lu-PSMA-617) that carries a radioactive component to destroy tumor cells. When lutetium is injected into the body, it attaches to the PSMA receptor found on tumor cells. After lutetium attaches to the PSMA receptor, its radiation component destroys the tumor cell. Giving 177Lu-PSMA-617 for 5 cycles versus 6 cycles may better treat patients with metastatic castrate resistant prostate cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine whether composite progression-free survival (PFS) per Prostate Cancer Clinical Trials Working Group 3 (PCWG3)-modified Response Evaluation Criteria in Solid Tumors (RECIST) 1.1, by physician discretion on prostate specific membrane antigen (PSMA)-positron emission tomography (PET), or biochemical progression is non-inferior among patients randomized to treatment pause versus standard treatment in patients with metastatic castrate resistant prostate cancer (mCRPC) who have minimal residual disease on post-therapy single photon emission computed tomography (SPECT) after 2 to 5 cycles of 177Lu-PSMA-617 treatment.

SECONDARY OBJECTIVES:

I. To compare time to subsequent treatment (TTST) in this patient population between randomized arms.

II. To assess time to radiographic progression per PCWG3-modified RECIST 1.1 or by physician discrection on PSMA PET between randomized arms in this patient population between randomized arms.

III. To assess overall survival (OS) in this patient population between randomized arms.

IV. To compare toxicities in treatment pause versus standard treatment in this patient population.

V. To assess changes in patient quality of life (QOL) as measured by the Functional Assessment of Cancer Therapy - Radionuclide Therapy (FACIT-RNT) for each randomized arm.

OUTLINE: Patients are randomized to 1 of 3 arms.

ARM I: Patients receive 177Lu-PSMA-617 intravenously (IV) over 10-15 minutes on day 1 of each cycle. Cycles repeat every 42 days for 5 cycles in the absence of disease progression or unacceptable toxicity. Patients with a near complete response may receive 1 additional cycle. Patients receive 68Ga-prostate specific membrane antigen-11 (gallium Ga 68-labeled PSMA-11) IV and undergo positron emission tomography (PET)/computed tomography (CT) during screening and on the trial. Patients also undergo SPECT/CT and blood sample collection on the trial.

ARM II: Patients receive 177Lu-PSMA-617 IV over 10-15 minutes on day 1 of each cycle. Cycles repeat every 42 days for 5 cycles in the absence of disease progression or unacceptable toxicity. Patients then undergo clinical observation until documented first progression. After progression, patients resume treatment with 77Lu-PSMA-617 for another cycle. Patients receive gallium Ga 68-labeled PSMA-11 IV and undergo PET/CT during screening and on the trial. Patients also undergo SPECT/CT and blood sample collection on the trial.

ARM III: Patients undergo clinical observation until documented first progression. After progression, patients receive 177Lu-PSMA-617 IV over 10-15 minutes on day 1 of each cycle. Cycles repeat every 42 days for 6 cycles in the absence of disease progression or unacceptable toxicity. Patients receive gallium Ga 68-labeled PSMA-11 IV and undergo PET/CT during screening and on the trial. Patients also undergo SPECT/CT and blood sample collection on the trial.

After completion of study treatment, patients are followed up every 12 weeks for up to 2 years or progressive disease.

ELIGIBILITY:
Inclusion Criteria:

* REGISTRATION INCLUSION CRITERIA
* Scheduled at Mayo Clinic Rochester for therapy with 177Lu PSMA-617
* PSMA positive metastatic castration resistant prostate cancer (68Ga and 18F PSMA PET will be considered equivalent for eligibility) , defined by molecular imaging prostate specific membrane antigen (miPSMA) score >= 2 on Mayo PET report, including interpretation of outside PET or consensus review of PET by nuclear therapy tumor board note in the patient chart
* Willingness to provide mandatory blood draws for correlative research. (This requirement is waived for patients enrolling after receiving cycle 1 of 177Lu PSMA-617,and achieving a near complete response on post therapy SPECT, as these patients will not be able to provide a pre-treatment baseline blood sample.)
* Provide written informed consent
* Ability to complete questionnaire(s) by themselves or with assistance
* Willing to return to enrolling institution for follow-up (during the active monitoring phase of the study)
* RANDOMIZATION INCLUSION CRITERIA
* Lesions with uptake equal to or above liver on cycle 1 post therapy SPECT, demonstrating that a near complete response on follow up post-therapy scan represents response, rather than sensitivity differences between SPECT and pre-treatment PET
* Near-complete response on post-therapy SPECT following any of cycles 2-5 of 177Lu PSMA-617. Near-complete response will be defined as no lesions with SUV max above the mean standard uptake value (SUV) of a representative 2cm spherical region of interest in the central right hepatic lobe, as determined by a nuclear medicine trained radiologist
* No toxicity that would indicate withholding or reducing dose of the next scheduled cycle of 177Lu PSMA-617 per prescribing information
* Hemoglobin (Hgb) ≥ 8 g/dL
* Platelets ≥ 75,000/mm^3
* Neutrophils ≥ 100/mm^3
* Estimated glomerular filtration rate (eGFR) < 50 mL/min *body surface area (BSA) using Cockcroft-Gault formula OR
* Creatinine ≤ 1.5 x upper limit of normal
* Aspartate transferase (AST) or alanine transaminase (ALT) ≤ 3 x upper limit of normal
* No other unacceptable toxicity in the clinical judgement of the investigators
* RE-REGISTRATION INCLUSION CRITERIA (CROSSOVER TO COMPLETION UPON FIRST PROGRESSION OF PATIENTS RANDOMIZED TO TREATMENT PAUSE)
* First progression in patients randomized to pause treatment
* PSMA avid lesions on PSMA PET (miPSMA score ≥ 2 following first progression)

Exclusion Criteria:

* REGISTRATION EXCLUSION CRITERIA
* Another active malignancy requiring therapy such as radiation, chemotherapy, or immunotherapy
* Receiving any other investigational agent which would be considered as a treatment for the prostate cancer
* Failure to recover from acute, reversible effects of prior therapy regardless of interval since last treatment

  * EXCEPTION: Grade 1 peripheral (sensory) neuropathy that has been stable for at least 3 months since completion of prior treatment
* Uncontrolled intercurrent non-cardiac illness including, but not limited to:

  * Ongoing or active infection
  * Psychiatric illness/social situations
  * Dyspnea at rest due to complications of advanced malignancy or other disease that requires continuous oxygen therapy
  * Any other conditions that would limit compliance with study requirements
* Any of the following because this study involves: An investigational agent whose genotoxic, mutagenic and teratogenic effects on the developing fetus and newborn are unknown

  * Persons able to father a child who are unwilling to employ adequate contraception
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* History of myocardial infarction ≤6 months, or congestive heart failure requiring use of ongoing maintenance therapy for life-threatening ventricular arrhythmias
* RE-REGISTRATION EXCLUSION CRITERIA
* Serious adverse effect

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 236 (Estimated)
Dates: Start 2024-05-03 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | Up to 5 years
  Progression free survival is defined as the time interval between randomization date and the date of disease progression or death, whichever occurs first. Progression will be defined in keeping with Prostate Cancer Clinical Trials Working Group 3 (PCWG3) guidelines. The median progression free survival of each arm, corresponding 95% confidence intervals, and hazard ratio comparing the treatment arm to the control arm will be reported.

SECONDARY OUTCOMES:
Time to subsequent treatment (TTST) | Up to 5 years
  TTST is defined as the time from randomization to subsequent treatment. Median TTST will be estimated using the Kaplan-Meier method. Patients who do not progress to a subsequent treatment while on study will be censored at the last known follow-up date. The median TTST and corresponding 95% confidence interval will be reported by randomized arm. The log-rank test will be used to compare the two arms on the distribution of TTST.
Time to progression (TTP) | Up to 5 years
  TTP is defined as the time from randomization to disease progression. Median TTP will be estimated using the Kaplan-Meier method. Patients who do not experience disease progression while on study will be censored at the last disease assessment date. Deaths will be censored. The median TTP and corresponding 95% confidence interval will be reported by randomized arm. The log-rank test will be used to compare the two arms on the distribution of TTP.
Overall survival (OS) | Up to 5 years
  Overall survival is defined as the time from study entry to death from any cause. Vital status and death dates will be obtained be electronic medical record review where possible, and by phone call where unavailable. Median OS will be estimated using the Kaplan-Meier method. Patients who do not experience death while on study will be censored at the last known date alive. The median OS and corresponding 95% confidence interval will be reported by randomized arm. The log-rank test will be used to compare the two arms on the distribution of OS.
Incidence of adverse events | Up to 5 years
  Adverse events will be summarized by frequency and severity using Common Terminology Criteria for Adverse Events (CTCAE) v 5.0. The proportion of patients who experience a grade 3+ adverse event at least possibly related to treatment will be reported by arm.
Quality of life - FACT-RNT | Up to 5 years
  Will be collected using the Functional Assessment of Cancer Therapy - Radionuclide Therapy (FACT-RNT). The FACT-RNT is a 15-item measure assessing symptoms and toxicities on a 0-4 scale. Total scores range from 0-60, with higher scores indicating better quality of life. Mean values at each collection timepoint will be plotted and stratified by randomized arm.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew P. Thorpe, M.D., Ph.D., Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials